CLINICAL TRIAL: NCT06588712
Title: Nutritional Assessment in Individuals with Liver Cirrhosis (Nutri-CIRR)
Brief Title: Nutritional Assessment in Individuals with Liver Cirrhosis
Acronym: Nutri-CIRR
Status: Not yet recruiting | Type: Observational
Sponsor: Université Sorbonne Paris Nord (Other)
Collaborators: Hôpital Henri Mondor, AP-HP, Unité de Recherche Clinique (Unknown); Hôpital Avicenne, AP-HP, Service Hépatologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-A01392-43
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with liver cirrhosis: Patients with liver cirrhosis are included in the cohort

SUMMARY:
The risk factors for liver cirrhosis are well identified and primarily include excessive and prolonged alcohol consumption, as well as metabolic syndrome or infection with hepatitis B and C viruses. However, the factors that can predict the progression of the disease are still largely unknown. The role of nutritional factors, in particular, has been insufficiently studied in chronic liver diseases such as cirrhosis. Beyond malnutrition and nutritional deficiencies, whose roles have been well studied, it appears that other nutritional factors, such as adherence to dietary recommendations that consider the consumption of various food groups, have been little studied in patients with liver cirrhosis. Studies involving a large number of participants are essential to better describe the typical nutritional profiles of these patients, taking into account their diet, as well as their alcohol consumption and physical activity.

Therefore, the main aim of the Nutri-CIRR project is to identify and characterize typical profiles of patients with hepatic cirrhosis in terms of nutritional factors (diet, alcohol consumption and physical activity) and smoking status.

DETAILED DESCRIPTION:
The Nutri-CIRR study is an observational study taking place in France and assessing nutritional factors among patients with liver cirrhosis. After inclusion in the study, all patients are invited to complete validated online questionnaires on diet, alcohol consumption, physical activity, as well as socioeconomic and other lifestyle characteristics. Questionnaires are completed at one occasion.

The main aim of the Nutri-CIRR project is to identify and characterize typical profiles of patients with hepatic cirrhosis in terms of nutritional factors (diet, alcohol consumption and physical activity) and smoking status.

Secondary aims are:

* Secondary aim #1: To describe values of the PNNS-GS2 score categorized into quantiles, which takes into account nutritional factors (diet, alcohol consumption and physical activity)
* Secondary aim #2: To evaluate the associations between nutritional factors (diet, alcohol consumption, physical activity) and the subsequent occurrence of hepatocellular carcinoma
* Secondary aim #3: To determine whether nutritional factors (diet, alcohol consumption, physical activity) are associated with competing hepatic risks (ascites, jaundice, bleeding due to portal hypertension, severe bacterial infections) and extra-hepatic risks (cardiovascular events, extra-hepatic cancers).

To address secondary aims #2 and #3, data from the Nutri-CIRR study will be matched with data from the FASTRAK study (NCT05095714), which monitors the liver disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Histologically proven cirrhosis or unequivocally suggested by non-invasive tests
* No HCC on imaging dated less than 3 months
* Ability to understand and read French, at the investigator's discretion
* Affiliation with a social security system

Exclusion Criteria:

* Child-Pugh C score
* Active hepatitis B or C
* Patient under legal protection
* Patient deprived of liberty
* Pregnant or breastfeeding woman, as known by the investigator
* Patient under State Medical Assistance (AME)
* Patient opposed to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Nutritional intakes | At enrollment
  Usual macronutrient and micronutrient intakes, assessed with a validated food frequency questionnaire
Food group intakes | At enrollment
  Usual intake of the main food groups, assessed with a validated food frequency questionnaire
Mediterranean diet score | At enrollment
  Mediterranean diet score, assessed with a validated food frequency questionnaire
Alcohol intake | At enrollment
  Usual alcohol intake, total and by type of alcoholic beverages, assessed with a validated food frequency questionnaire
Smoking status | At enrollment
  Smoking status, number of pack-years, assessed by questionnaire
Physical activity | At enrollment
  Duration of moderate and vigorous physical activity, duration of walking, physical activity level (low, moderate, high, calculated using the duration of moderate, vigorous physical activity and walking), assessed with the IPAQ short-form
Sedentary behavior | At enrollment
  Sitting time, assessed with the IPAQ short-form
Weight | At enrollment
  Self-reported body weight
Height | At enrollment
  Self-reported height
Body mass index | At enrollment
  Calculated as weight/(height*height)
Nutritional score | At enrollment
  PNNS-GS2 is a nutritional score calculated using data on dietary intake, alcohol intake and physical activity. A higher score indicates a greater nutritional quality

SECONDARY OUTCOMES:
Socioeconomic factors | At enrollment
  Educational, level, occupation, income
Demographic factors | At enrollment
  Gender, marital status, household composition, number of children
Follow-up of cirrhotic disease (occurrence of hepatocellular carcinoma) | From enrollment to the end of follow-up at 3 years
  Occurrence of hepatocellular carcinoma. These data will be collected as part of a matching process with the FASTRAK study (NCT05095714) for patients included in both studies (Nutri-CIRR + FASTRAK)
Follow-up of cirrhotic disease (other hepatic complications) | From enrollment to the end of follow-up at 3 years
  Occurrence of other hepatic complications (ascites, jaundice, bleeding due to portal hypertension, severe bacterial infections). These data will be collected as part of a matching process with the FASTRAK study (NCT05095714) for patients included in both studies (Nutri-CIRR + FASTRAK)
Follow-up of cirrhotic disease (extra-hepatic complications) | From enrollment to the end of follow-up at 3 years
  Occurrence of extra-hepatic complications (cardiovascular events, extra-hepatic cancers). These data will be collected as part of a matching process with the FASTRAK study (NCT05095714) for patients included in both studies (Nutri-CIRR + FASTRAK)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bellicha, PhD, Principal Investigator — Université Sorbonne Paris Nord

IPD SHARING:
Plan to Share IPD: Undecided
Data described in the article, code book, and analytic code will be made available upon request. Researchers of a public institution can submit a collaboration request including their institution and a brief description of their project to the principal investigator. All requests will be reviewed by the scientific team of the project. A financial contribution may be requested. If the collaboration is accepted, a data access agreement will be necessary and appropriate authorizations from the competent administrative authorities may be needed. In accordance with existing regulations, no personal data will be accessible.